CLINICAL TRIAL: NCT05735548
Title: Prognostic Factors in Tumors of the Peripheral Nervous System
Brief Title: Tumors of the Peripheral Nervous System
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: ID 3787
Record Dates: First submitted 2023-01-31; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Tumor of Peripheral Nerve
Keywords: outcome, neurosurgery
MeSH Terms: conditions — Peripheral Nervous System Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to individuate tumors' and patients' features influencing the outcome after surgical tumor removal.

DETAILED DESCRIPTION:
Patients operated because of removal of Peripheral Nervous System (PNS) tumor will be recruited accordingly to the inclusion criteria: the aims of the study will be illustrated and the informed consent signed.

All the clinical and neuroradiological perioperative documents of the enrolled patients will be analyzed. As follow-up, thorough neurological exam wil be performed and specific surveys about after surgery social and working life will be administered; neuroradiological imaging will be performed.

Then, the results will be investigated to individuate which factors were related to the outcome.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 y.o.
* neurosurgical removal of peripheral nerve tumor at our University Hospital "Fondazione Policlinico Universitario Agostino Gemelli (FPG)" during the previous 10 years
* signed consent to study participation

Exclusion Criteria:

* < 18 y.o.
* neurosurgical treatment because other causes (chronic entrapment syndromes, acute nerve lesion)
* denied consent to study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed histology of peripheral nerve tumor, operated at our hospital during the 10 years before the study started.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
oncological outcome | through study completion, an average of 3 years
  number of patients with tumor relapses
functional outcome | through study completion, an average of 3 years
  evaluation of: 1) Motor function accordingly to the "Medical Research Council muscle power scale (MRC); 2) Sensation accordingly to "The Ten Test for Sensation" (TTTS); 3) Pain accordingly to the "Numerical Rating Scale for Pain" (NRS).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy